CLINICAL TRIAL: NCT07197424
Title: Robot Assisted Magnetically Controlled Capsule Endoscopy
Brief Title: The Use of Robot Assisted Magnetically Controlled Capsule Endoscopy in Patients With Iron Deficiency Anaemia
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: University of Edinburgh (Other)
Collaborators: NHS Lothian (Other Government)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Other
Other Study IDs: REC Number: 25/YH/0132; Sponsor number: AC25074 (Other: University of Edinburgh); IRAS Study ID: 349888 (Other: IRAS); R&D Number: 2025/0152 (Other: NHS Lothian)
Record Dates: First submitted 2025-09-18; First posted 2025-09-29 (Actual); Last update posted 2025-11-25 (Actual); Status verified 2025-08

CONDITIONS: Iron Deficiency Anaemia
Keywords: capsule endoscopy; robot assisted magnetically controlled capsule endoscopy; iron deficiency anaemia
MeSH Terms: conditions — Anemia, Iron-Deficiency | interventions — Endoscopy

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Robot assisted magnetically controlled capsule endoscopy (Other)
  Interventions: Diagnostic Test: Robot assisted magnetically controlled capsule endoscopy

INTERVENTIONS:
Diagnostic Test: Robot assisted magnetically controlled capsule endoscopy — Examination of the upper GI tract (oesophagus and stomach) with robot assisted magnetically controlled capsule endoscopy. Examination of the small bowel will be completed using the same capsule, however it will not be robot assisted.

SUMMARY:
In this study the investigators will recruit patients who have already had an upper gastrointestinal (GI) tract endoscopy (OGD) and lower GI tract investigations which did not identify the source of iron deficiency anaemia, and who need the small bowel to be investigated. This will comprise both patients who would have proceeded directly to small bowel capsule endoscopy (SBCE) under standard care and also those from whom an initial 'watch and wait' approach may have been adopted before proceeding to SBCE. The investigators propose to investigate these patients during a single patient visit to Leith Community Treatment Centre, Edinburgh, Scotland, with a CE marked robotic capsule system which can examine both the upper GI tract (i.e. the oesophagus and the stomach) and the small bowel in one investigation using a magnetic guided capsule.

The aim of the study is to compare the findings from OGD with the robotic capsule system and to determine if such a system may safely replace OGD - thus examining the upper GI tract and small bowel for IDA in one less invasive investigation. This has the potential to decrease patient discomfort, stress and anxiety, while also reducing pressure on busy endoscopy departments, helping to ensure that the right patients receive the right investigations in a timely manner.

ELIGIBILITY:
Inclusion Criteria:

* Adult patients aged 18 and above
* Confirmed diagnosis of iron deficiency anaemia (either recent onset or recurrent)
* No significant cause for iron deficiency anaemia previously identified on upper GI endoscopy, colonoscopy or CT colonography
* Patients who would either have proceeded directly to small bowel capsule endoscopy (SBCE) or who would have had an initial 'watch and wait' period prior to undergoing SBCE

Exclusion Criteria:

* Known or suspected gastrointestinal obstruction, strictures or fistulae
* Previous abdominal surgery
* Dysphagia
* Patients with a pacemaker, defibrillator or other implanted electronic device
* In vivo retention with medical metal fittings - shunts, plates, stents or clips
* A history of metal fragments in the eyes or elsewhere in the body
* Confirmed or possible pregnancy
* Patients who are not deemed to have capacity according to the Adults with Incapacity Act
* Patients who are currently part of another research study

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 100 (Estimated)
Dates: Start 2025-12-31 (Estimated); Primary Completion 2027-03 (Estimated); Study Completion 2027-03 (Estimated)

PRIMARY OUTCOMES:
Non-inferiority of robot assisted magnetically controlled capsule endoscopy compared to upper GI endoscopy (OGD) | From individual patient enrolment to completion and reporting of capsule endoscopy examination
  The principal research objective that this study seeks to address is if robot assisted magnetically controlled capsule endoscopy may be safely and effectively used as an alternative to upper GI endoscopy (OGD) (i.e. it is non-inferior when compared to OGD) in the investigation of patients with iron deficiency anaemia.
  This will be achieved through a review of OGD reports, the findings of which will be recorded. These will be directly compared to the findings at robot assisted magnetically controlled capsule endoscopy and any differences noted. Cohen's kappa coefficient will be used to assess the degree of diagnostic agreement between OGD and robot assisted magnetically controlled capsule endoscopy, with reference to the total number of lesions and specific pathology detected.

CONTACTS AND LOCATIONS:
Overall Officials: John N Plevris, MD, DM, PhD(E), FRCPE, FEBGH, Principal Investigator — University of Edinburgh
Locations (1):
- Leith Community Treatment Centre, Edinburgh, United Kingdom

IPD SHARING:
Plan to Share IPD: No
Data will not be shared at an individual patient level

REFERENCES:
- [Background] Xiao YF, Wu ZX, He S, Zhou YY, Zhao YB, He JL, Peng X, Yang ZX, Lv QJ, Yang H, Bai JY, Fan CQ, Tang B, Hu CJ, Jie MM, Liu E, Lin H, Koulaouzidis A, Zhao XY, Yang SM, Xie X. Fully automated magnetically controlled capsule endoscopy for examination of the stomach and small bowel: a prospective, feasibility, two-centre study. Lancet Gastroenterol Hepatol. 2021 Nov;6(11):914-921. doi: 10.1016/S2468-1253(21)00274-0. Epub 2021 Sep 21. PMID 34555347